CLINICAL TRIAL: NCT00949364
Title: Multi-Center Phase II Study With Pomalidomide in Patients With Myeloproliferative Neoplasms in Fibrotic Stage
Brief Title: Pomalidomide in Patients With Myeloproliferative Neoplasms in Fibrotic Stage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard Schlenk, Prof.Dr., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPN-SG 01-09
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Myeloproliferative Neoplasms; Pomalidomide; Fibrotic Stage; Patients with Myeloproliferative Neoplasms in Fibrotic Stage
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide (Experimental): Every patient will remain on treatment until disease progression for at least 12 cycles, withdrawal of patient's informed consent or the occurrence of unacceptable toxicity. If a patient may benefit from treatment with pomalidomide the investigator together with the principle investigator will discuss the possibility of further treatment including maintenance treatment with pomalidomide on a case-by-case decision. This additional treatment will be performed within the follow-up period of the study, data will be collected and duration will be maximally 12 cycles.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Treatment starts with pomalidomide as single agent therapy: 0.5 mg/day. Prednisolone will be started in the absence of PD as randomized either at start of cycle 4 or start of cycle 7 (starting dose: 30 mg/day for 28 days followed by 15 mg/day and 10 mg/day for 28 days), if no response acc. to IWG-MRT (no CR, PR, CI, TI) was achieved.
  If PD: treatment is stopped. Otherwise, continuous treatment at least until end of cycle 12 is intended. For patients responding to the combination treatment (pomalidomide/prednisolone) a concom. treatment after cycle 6 or 9 (depending on the randomization result) with prednisolone in doses equal or below 7.5 mg/day are allowed.
  If a patient may benefit from treatment with pomalidomide the invest. and the PI will discuss the possibility of further treatment including maintenance treatment with pomalidomide on a case-by-case decision (max. duration: 12 cycles).

SUMMARY:
This is a phase II, multi-center study of pomalidomide in adult patients with PMF, SMF, and unclassifiable MPN showing at least grade 1 bone marrow fibrosis and requiring therapy. All patients will receive per oral pomalidomide on a daily basis.

First cohort (Before Amendment No. 1 ID 1-41):

Treatment starts with a phase of pomalidomide therapy with 2 mg per day. Individual dose reduction as outlined in the safety section is allowed. If no response was achieved (no complete remission (CR), partial response (PR), clinical improvement (CI) and no progressive disease according to the IWG-MRT criteria) after 3 months, prednisolone is added in a starting dose of 30 mg per day. In the absence of progressive disease, at least 6 months of treatment with pomalidomide is intended. In patients without disease progression after 6 months and those with response to treatment are intended to receive pomalidomide for at least 12 months. Additional antiproliferative treatment with hydroxyurea for leukocytosis (>20 x 109/l) and/or thrombocytosis (>750 x 109/l) and/or symptomatic splenomegaly in a starting dose of 2g/day with individual dose adjustment is allowed.

Second cohort (After Amendment No. 1 ID > 41):

To evaluate the relative impact of prednisolone to the objective response rate, a randomization has been integrated into the study concept. The addition of prednisolone is up-front randomized for the start of prednisolone either after 3 or 6 cycles of treatment with pomalidomide as single agent if no response occurred during this period. This results in the following treatment arms:

Treatment Arm A) Pomalidomide 0.5 mg per day + additional prednisolone at start of cycle 4 (day 85), in case no response was achieved until end of cycle 3.

Treatment Arm B) Pomalidomide 0.5 mg per day + additional prednisolone at start of cycle 7 (day 169), if no response was achieved until end of cycle 6.

Treatment for all patients starts with pomalidomide as single agent at a dose of 0.5mg per day. The addition of prednisolone will be initiated as randomized either at start of cycle 4 or start of cycle 7 (starting dose 30 mg per day). In the absence of progressive disease, at least 12 cycles of treatment with pomalidomide are intended.

Additional antiproliferative treatment with hydroxyurea for leukocytosis (>20 x 109/l) and/or thrombocytosis (>750 x 109/l) and/or symptomatic splenomegaly in a starting dose of 2g/day with individual dose adjustment is allowed.

ELIGIBILITY:
Inclusion Criteria:

Both female and male patients meeting the mentioned inclusion and exclusion criteria will be included in this clinical trial. The risk to get PMF or SMF does not depend on a patient's gender. Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Age ≥50 years at the time of voluntarily signing an IRB/IEC-approved informed consent
2. Diagnosis of Myeloproliferative Neoplasms (MPN) either de novo myelofibrosis according to WHO criteria (PMF) [20], secondary myelofibrosis (post-PV MF and post-ET MF according to the IWG-MRT consensus terminology) [21] or unclassifiable MPN with biopsy proven myelofibrosis
3. Anemia with hemoglobin level of <10 g/dl or transfusion-dependent anemia and/or thrombocytopenia <50 /nl or transfusion-dependent thrombocytopenia and/or neutropenia <1.0 /nl
4. Splenomegaly (>11 cm diameter) and/or leukoerythroblastosis
5. Adequate organ function, i.e. ALT and/or AST <3 x upper limit of normal (ULN), total bilirubin <3 x ULN, and serum creatinine <2 mg/dl
6. Subject must be willing to receive transfusion of blood products
7. ECOG performance status < 3
8. Female subjects with non-childbearing potential:

   * Agree to have a pregnancy test at baseline
9. Male subjects:

   * Agree to use condoms throughout study drug therapy, during any dose interruption and for four weeks after cessation of study therapy if their partner is of childbearing potential and has no contraception.
   * Agree not to donate semen during study drug therapy and for four weeks after end of study drug therapy.
10. All Subjects:

    * Will be counseled about potential teratogenic risks of the study medication.
    * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
    * Agree not to share study medication with another person and to return all unused study drug to the investigator
    * No more than a 12-weeks-supply of study drug will be dispensed at a time.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Females of childbearing potentials°, pregnant or breast feeding females
2. BCR/ABL-positivity
3. Diagnosis of ET (according to WHO 2008 criteria)
4. Diagnosis of PV (according to WHO 2008 criteria)
5. >20% blasts in peripheral blood or bone marrow
6. Known positive status for HIV, HBV or HCV
7. Prior treatment with IMiDs (thalidomide, lenalidomide) or with Interferon-alpha within a 3 month time period before screening
8. History of thrombosis or pulmonary embolism
9. Peripheral neuropathy >grade 1 CTC
10. No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.
11. Presence of any medical/psychiatric condition or laboratory abnormalities which may limit full compliance with the study, increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
12. Drug or alcohol abuse within the last 6 months
13. Patients with a "currently active" second malignancy other than nonmelanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.

Criteria for women of non-childbearing potential:

A female patient or a female partner of a male patient is considered to have childbearing potential unless she meets at least one of the following criteria:

* Age ≥ 50 years and naturally amenorrhoeic for ≥ 1 year. Amenorrhoea following cancer therapy does not rule out childbearing potential
* Premature ovarian failure confirmed by a specialist gynecologist
* Previous bilateral salpingo-oophorectomy, or hysterectomy
* XY genotype, Turner syndrome, uterine agenesis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-12; Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Objective disease response, as defined by the IWG-MRT criteria for response in MF patients extended by the criterion RBC-transfusion independence (TI) | one year

SECONDARY OUTCOMES:
Overall safety profile of pomalidomide characterized by type, frequency, severity, timing and relatedness of adverse events (AEs) and laboratory abnormalities observed during treatment | one year
  Graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 3.0
Event-free survival | three years
Relapse-free survival | three years
Overall survival | three years

CONTACTS AND LOCATIONS:
Locations (15):
- Germany (15):
  - Universitätsklinikum Aachen, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - Zentrum für Ambulante Hämatologie und Onkologie, Bonn
  - BAG Freiberg-Richter, Jacobasch, Wolf, Illmer (Gemeinschaftspraxis), Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum der Johann Goethe-Universität Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg Eppendorf, Hamburg Eppendorf
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Haematologisch-onkologische Praxis, München
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Result] Schlenk RF, Stegelmann F, Reiter A, Jost E, Gattermann N, Hebart H, Waller C, Hochhaus A, Platzbecker U, Schafhausen P, Blau IW, Verbeek W, Heidel FH, Werner M, Kreipe H, Teleanu V, Benner A, Dohner H, Griesshammer M, Dohner K. Pomalidomide in myeloproliferative neoplasm-associated myelofibrosis. Leukemia. 2017 Apr;31(4):889-895. doi: 10.1038/leu.2016.299. Epub 2016 Oct 24. PMID 27774990